CLINICAL TRIAL: NCT04085523
Title: ACcomplisH: A Phase 2, Multicenter, Double-blind, Randomized, Placebo-controlled, Dose Escalation Trial Evaluating Safety, Efficacy, and Pharmacokinetics of Subcutaneous Doses of TransCon CNP Administered Once Weekly for 52 Weeks in Prepubertal Children With Achondroplasia Followed by an Open-Label Extension Period
Brief Title: A Dose Escalation Trial Evaluating Safety, Efficacy, and Pharmacokinetics of TransCon CNP Administered Once Weekly in Prepubertal Children With Achondroplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascendis Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCC-201
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Results first posted 2024-03-07 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Achondroplasia
Keywords: Achondroplasia; Dwarfism
MeSH Terms: conditions — Achondroplasia; Dwarfism

STUDY DESIGN:
Intervention Model Description: There are 5 cohorts enrolling approximately 60 subjects who will be randomized to receive either TransCon CNP or Placebo in a 3:1 ratio
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- TransCon CNP 6 mcg (Experimental): TransCon CNP 6 mcg CNP/kg delivered once weekly by subcutaneous injection.
  Interventions: Drug: TransCon CNP
- TransCon CNP 20 mcg (Experimental): TransCon CNP 20 mcg CNP/kg delivered once weekly by subcutaneous injection.
  Interventions: Drug: TransCon CNP
- TransCon CNP 50 mcg (Experimental): TransCon CNP 50 mcg CNP/kg delivered once weekly by subcutaneous injection.
  Interventions: Drug: TransCon CNP
- TransCon CNP 100 mcg (Experimental): TransCon CNP 100 mcg CNP/kg delivered once weekly by subcutaneous injection.
  Interventions: Drug: TransCon CNP
- Placebo (Placebo Comparator): Placebo mimicking 6, 20, 50, or 100 mcg CNP/kg delivered once weekly by subcutaneous injection.
  Interventions: Drug: Placebo for TransCon CNP
- Open-Label Extension Period: TransCon CNP (Experimental): Participants who completed the 52-week blinded treatment period continued into the 104-week open-label extension period and received treatment with TransCon CNP (navepegritide) doses escalated up to a maximum of 100 mcg/kg delivered once weekly by subcutaneous injection.
  Interventions: Drug: TransCon CNP

INTERVENTIONS:
Drug: TransCon CNP — TransCon CNP drug product is a lyophilized powder in a single-use vial containing either TransCon CNP 3.9 mg CNP-38/vial or TransCon CNP 0.80 mg CNP-38/vial. Prior to use, the lyophilized powder is reconstituted with sterile water for injection and administered by subcutaneous injection via syringe and needle.
  Arms: Open-Label Extension Period: TransCon CNP; TransCon CNP 100 mcg; TransCon CNP 20 mcg; TransCon CNP 50 mcg; TransCon CNP 6 mcg
Drug: Placebo for TransCon CNP — Weekly subcutaneously injection of placebo.
  Arms: Placebo

SUMMARY:
The trial is a multicenter, double-blind, randomized, placebo-controlled, dose escalation trial of weekly TransCon CNP administered subcutaneously in prepubertal children 2 to 10 years old, inclusive, with Achondroplasia.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of ACH with genetic confirmation
2. Age between 2 to 10 years old (inclusive) at Screening Visit
3. Prepubertal (Stage 1 breasts for girls or testicular volume < 4ml for boys) at Screening Visit
4. Able to stand without assistance
5. Caregiver willing and able to administer subcutaneous injections of study drug

Exclusion Criteria:

1. Clinically significant findings at Screening that:

   * are expected to require surgical intervention during participation in the trial or
   * are musculoskeletal in nature, such as Salter-Harris fractures and severe hip pain or
   * otherwise are considered by investigator or Medical Monitor/Medical Expert to make a participant unfit to receive study drug or undergo trial related procedures
2. Have received treatment (>3 months) of human growth hormone (hGH) or other medications known to affect stature or body proportionality at any time
3. Have received any dose of medications intended to affect stature or body proportionality within the previous 6 months of Screening Visit
4. Have received any study drug or device intended to affect stature or body proportionality at any time
5. History or presence of injury or disease of the growth plate(s), other than Achondroplasia, that affects growth potential of long bones

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee D. Shu, MD, Study Director — Ascendis Pharma, Inc.
Locations (15):
- United States (8):
  - Ascendis Pharma Investigational Site, Little Rock, Arkansas
  - Ascendis Pharma Investigational Site, Aurora, Colorado
  - Ascendis Pharma Investigational Site, Saint Paul, Minnesota
  - Ascendis Pharma Investigational Site, Columbia, Missouri
  - Ascendis Pharma Investigational Site, Buffalo, New York
  - Ascendis Pharma Investigational Site, Houston, Texas
  - Ascendis Pharma Investigational Site, Seattle, Washington
  - Ascendis Pharma Investigational Site, Madison, Wisconsin
- Ascendis Pharma Investigational Site, Parkville, Victoria, Australia
- Ascendis Pharma Investigational Site, Linz, Austria
- Ascendis Pharma Investigational Site, Copenhagen, Denmark
- Ascendis Pharma Investigational Site, Berlin, Germany
- Ascendis Pharma Investigational Site, Dublin, Ireland
- Ascendis Pharma Investigational Site, Auckland, New Zealand
- Ascendis Pharma Investigational Site, Coimbra, Portugal

REFERENCES:
- [Result] Savarirayan R, Hoernschemeyer DG, Ljungberg M, Zarate YA, Bacino CA, Bober MB, Legare JM, Hogler W, Quattrin T, Abuzzahab MJ, Hofman PL, White KK, Ma NS, Schnabel D, Sousa SB, Mao M, Smith A, Chakraborty M, Giwa A, Winding B, Volck B, Shu AD, McDonnell C. Once-weekly TransCon CNP (navepegritide) in children with achondroplasia (ACcomplisH): a phase 2, multicentre, randomised, double-blind, placebo-controlled, dose-escalation trial. EClinicalMedicine. 2023 Oct 2;65:102258. doi: 10.1016/j.eclinm.2023.102258. eCollection 2023 Nov. PMID 37823031

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 60 participants were screened and 57 participants met eligibility criteria and were enrolled into the trial and randomized in the planned ratio of approximately 3:1 (TransCon CNP: Placebo) within sequential dose escalation cohorts. All 57 participants completed the 52-week double-blind period & entered the 104-week open-label extension (OLE) period, where they received TransCon CNP. All participants received up to a maximum of 100-mcg dose of TransCon CNP during the OLE period.
Period: Double-Blind Period (Weeks 0 to 52)
Arm/Group | TransCon CNP 6 mcg | TransCon CNP 20 mcg | TransCon CNP 50 mcg | TransCon CNP 100 mcg | Placebo | Open-Label Extension Period: TransCon CNP
Started | 10 | 11 | 10 | 11 | 15 | 0
Completed | 10 | 11 | 10 | 11 | 15 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Open-Label Period (Weeks 52 to 156)
Arm/Group | TransCon CNP 6 mcg | TransCon CNP 20 mcg | TransCon CNP 50 mcg | TransCon CNP 100 mcg | Placebo | Open-Label Extension Period: TransCon CNP
Started | 0 | 0 | 0 | 0 | 0 | 57 (Participants who completed the 52-week double blind treatment period.)
Completed | 0 | 0 | 0 | 0 | 0 | 55
Not Completed | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TransCon CNP 6 mcg | TransCon CNP 20 mcg | TransCon CNP 50 mcg | TransCon CNP 100 mcg | Placebo | Total
Number analyzed (Participants) | 10 | 11 | 10 | 11 | 15 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.52 (2.593) | 6.29 (2.896) | 5.20 (2.991) | 5.79 (2.613) | 5.89 (3.109) | 5.94 (2.800)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 3 | 6 | 5 | 24
  Male | 3 | 8 | 7 | 5 | 10 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 2 | 1 | 6
  Not Hispanic or Latino | 9 | 11 | 6 | 9 | 14 | 49
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 0 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 1 | 1 | 2
  White | 8 | 10 | 8 | 10 | 12 | 48
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 90.63 (8.973) | 92.29 (12.103) | 86.61 (12.967) | 89.23 (12.822) | 90.85 (14.920) | 90.03 (12.434)
Height SDS [Mean (Standard Deviation); unit: standard deviation score] — Height expressed in Standard Deviation Score (SDS) is derived using CDC 2000 (USA)/Kuczmarski method. A Height SDS of 0 represents the population mean or average. A lower SDS means the value is closer to the average and a higher SDS means the value is further from the average. A negative SDS indicates below average height and a positive SDS indicates above average height.
  standard deviation score | -5.45 (1.046) | -4.87 (0.673) | -4.85 (0.801) | -4.92 (0.829) | -4.85 (0.958) | -4.97 (0.873)
Weight [Mean (Standard Deviation); unit: kg] | 17.49 (3.677) | 19.67 (6.602) | 15.67 (4.399) | 17.03 (4.699) | 17.99 (5.542) | 17.64 (5.129)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 21.10 (1.664) | 22.52 (2.599) | 20.61 (1.496) | 21.11 (1.612) | 21.39 (1.853) | 21.36 (1.930)

OUTCOME MEASURES:

1. Primary Outcome: Annualized Height Velocity (cm/Year) After 52 Weeks of Double-blind Treatment
Description: The primary efficacy analysis compared the difference in the primary efficacy endpoint between the TransCon CNP treatment group and the pooled placebo group using an ANCOVA model with the annualized height velocity (AHV) at Week 52 as the response variable, treatment (dose groups and placebo) and sex as factors, baseline age and baseline height SDS as the covariates, and based on the Full Analysis Set.
Time Frame: 52 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: cm/year
Arm/Group | TransCon CNP 6 mcg | TransCon CNP 20 mcg | TransCon CNP 50 mcg | TransCon CNP 100 mcg | Placebo
Number analyzed (Participants) | 10 | 11 | 10 | 11 | 15
cm/year | 4.09 [3.34 to 4.84] | 4.52 [3.82 to 5.22] | 5.16 [4.43 to 5.90] | 5.42 [4.74 to 6.11] | 4.35 [3.75 to 4.94]
Statistical Analysis 1: Comparison: TransCon CNP 6 mcg vs Placebo; ANCOVA model using treatment (dose groups and pooled placebo) and sex as fixed effects, and baseline age and baseline height SDS as the covariates; Test type: Superiority; p = 0.6004, ANCOVA
Statistical Analysis 2: Comparison: TransCon CNP 20 mcg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.7022, ANCOVA
Statistical Analysis 3: Comparison: TransCon CNP 50 mcg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0849, ANCOVA
Statistical Analysis 4: Comparison: TransCon CNP 100 mcg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0218, ANCOVA

ADVERSE EVENTS:
Time Frame: From Week 0 to Week 52 for double-blind treatment period and up to Week 156 for OLE Period
Description: Analysis was performed on safety analysis set that included all randomized participants who received at least one dose of trial drug. Participants were analyzed according to trial treatment as treated. Adverse Events were reported as per MedDRA version 24.1 for double-blind treatment period and MedDRA version 26.0 for OLE period.
Arm/Group | TransCon CNP 6 mcg | TransCon CNP 20 mcg | TransCon CNP 50 mcg | TransCon CNP 100 mcg | Placebo | Open-Label Extension Period: TransCon CNP
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11 | 0/10 | 0/11 | 0/15 | 0/57
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/11 | 1/10 | 0/11 | 0/15 | 2/57
Other Adverse Events (participants affected / at risk) | 9/10 | 11/11 | 10/10 | 10/11 | 14/15 | 57/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TransCon CNP 6 mcg (N=10) | TransCon CNP 20 mcg (N=11) | TransCon CNP 50 mcg (N=10) | TransCon CNP 100 mcg (N=11) | Placebo (N=15) | Open-Label Extension Period: TransCon CNP (N=57)
Febrile Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TransCon CNP 6 mcg (N=10) | TransCon CNP 20 mcg (N=11) | TransCon CNP 50 mcg (N=10) | TransCon CNP 100 mcg (N=11) | Placebo (N=15) | Open-Label Extension Period: TransCon CNP (N=57)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 2 (8) | 17 (40)
Pyrexia (General disorders) | 1 (2) | 4 (7) | 2 (2) | 2 (4) | 5 (8) | 23 (56)
Injection Site Reaction (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 5 (24)
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 10 (22)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (4) | 2 (3) | 3 (3) | 3 (5) | 16 (25)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (2) | 2 (2) | 6 (8)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 4 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 3 (7) | 4 (6) | 2 (4) | 3 (5) | 21 (51)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (4) | 2 (2) | 1 (1) | 11 (18)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 2 (3) | 0 (0) | 3 (5) | 13 (31)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 10 (14)
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 7 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (7) | 3 (3) | 1 (1) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 1 (18) | 9 (14)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 5 (8) | 0 (0) | 2 (2) | 14 (22)
Nasopharyngitis (Infections and infestations) | 1 (2) | 0 (0) | 5 (6) | 2 (2) | 1 (3) | 20 (35)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 10 (13)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 20 (22)
Otitis media (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 14 (18)
Viral infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (4) | 0 (0) | 2 (3) | 8 (17)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 14 (27)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (10)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 7 (11)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 7 (15)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (6)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (8)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 4 (4)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (26)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (6)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (10)
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (10)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (7)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 5 (6)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 6 (8)
Vitamin D decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT04085523/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT04085523/SAP_001.pdf